CLINICAL TRIAL: NCT02298582
Title: Safety of Intranasal Fentanyl (PecFent®) in the Treatment of Procedural Pain in the Elderly With or Without Background Treatment.
Brief Title: Safety of Intranasal Fentanyl (PecFent®) in the Treatment of Procedural Pain in the Elderly
Acronym: FENTA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCIC/13/67
Record Dates: First submitted 2014-10-13; First posted 2014-11-24 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Pain Due to Certain Specified Procedures
Keywords: safety; procedural pain; intranasal fentanyl; elderly
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intranasal fentanyl (Experimental)
  Interventions: Drug: intranasal fentanyl

INTERVENTIONS:
Drug: intranasal fentanyl — During the two first sessions of care or rehabilitation, patients do not receive Pecfent® in order to assess their basal pain. During the following four sessions, patients will receive transmucosal fentanyl, 10 minutes before care. A titration of PecFent will be done at each session

SUMMARY:
The purpose of this study is to evaluate the safety of the intranasal fentanyl in pain induced by wound care and rehabilitation in the elderly. The project would also provide a preliminary assessment of the effectiveness of intranasal fentanyl used in procedural pains.

DETAILED DESCRIPTION:
This is a safety clinical trial. This trial is monocentric, open label, non-randomized.

Sixty elderly patients will be enrolled in this study, 30 with bedsore cares and 30 with rehabilitation sessions.

Six bedsore cares or rehabilitation sessions will be assessed for each subject. For each session, patient pain will be evaluated using a visual analogic scale VAS at different times, before session, 5 minutes then 20 minutes after the beginning of the session, and a last VAS 1 hour after the end of the session. During the two first sessions, patients do not receive Pecfent® to assess their basal pain. During the following four sessions, patients will receive transmucosal fentanyl, 10 minutes before care.

An evaluation of respiratory rate and of the level of sedation will occur at different time : after 5 minutes then 20 minutes of care, at the end of the care session,at half an hour then one hour after the care session.

At the end of sessions,

* The nurse or physiotherapist will assess their satisfaction regarding the objectives achieved during the session with a four points verbal descriptor scale (very satisfied, satisfied, not much satisfied, not satisfied). They will also evaluate at the end of the four last session their satisfaction regarding the convenience of the use of pecfent® and its contribution towards care.
* Patients will assess their satisfaction regarding the course of the session with a verbal descriptor scale (VDS) and their level of anxiety felt during the session with a VAS.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized geriatric patient requiring care or rehabilitation
* Patient with pain during treatment or mobilization. (VAS ≥ 4)
* Written Informed consent

Exclusion Criteria:

* All unstable fractures
* Confusion: unable to assess their level of pain using a VAS.
* Contraindications to PecFent ® (. Hypersensitivity to the active substance or to any of the excipients listed in section Composition Use in patients who had never received treatment for opioid severe respiratory depression or severe obstructive pulmonary disease.)
* Person under legal protection

Min Age: 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-12-08 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Safety of intranasal fentanyl as measured by the nature and frequency of adverse effects. | 5 days after the last intake of fentanyl.
  The nature and frequency of adverse effects will be described. The collection of adverse events will be first, with the collection of spontaneous patient complaints from nurses on the other hand, by systematic screening with the patient. Monitoring of respiratory rate and level of sedation will also be set up.

SECONDARY OUTCOMES:
Effectiveness of intranasal fentanyl in procedural pain using a VAS (Visual Analogic Scale) of pain. | Evolution of the level of pain (VAS) since the beginning of care until one hour after the end of session (on average at 2 hours).
  VAS will be evaluated during each session at t0, t0+15min, t0+30min, and 1hour after the session (on average at 2 hours)
Fentanyl impact on the goals of care as measured by a caregiver satisfaction scale. | At the end of session of care or rehabilitation (on average at 1 hour).
  At the end of each session of care or rehabilitation, it will be proposed to the caregiver, a scale measuring its satisfaction regarding the objectives achieved during the session.
Nurse or physiotherapist satisfaction regarding use of PecFent® as measured by a verbal descriptor scale | 1 hour after the last intake of fentanyl
  Nurse or physiotherapist evaluation satisfaction regarding the convenience of the use of pecfent® and its contribution towards care using a verbal descriptor scale
Impact of PecFent® on patient feelings during care or rehabilitation sessions as measured by a verbal descriptor scale | At the end of Session of care or rehabilitation (on average at 1 hour).
  Patient evaluation at the end of sessions:
  - Patient satisfaction regarding the course of the session with a VDS

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Grenoble, Grenoble, Isere, France